CLINICAL TRIAL: NCT03372447
Title: Megadose of Hydroxocobalamin (Vitamin B12) for the Treatment of Pernicious Anemia
Brief Title: Megadose of Hydroxocobalamin for the Treatment of Pernicious Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Principal Investigator / Head of Hematology Department/MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE17-00023
Record Dates: First submitted 2017-12-05; First posted 2017-12-13 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Megaloblastic Anemia Nos; Pernicious Anemia
MeSH Terms: conditions — Anemia, Megaloblastic; Anemia, Pernicious | interventions — Hydroxocobalamin; Thiamine; Pyridoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Megadose multivitamin complex (Experimental): Intramuscular injection of hydroxocobalamin 10,000mcg, Thiamin 100mg, Pyridoxine 50mg
  Interventions: Drug: Hydroxocobalamin 10,000mcg, Thiamin 100mg, Pyridoxine 50mg

INTERVENTIONS:
Drug: Hydroxocobalamin 10,000mcg, Thiamin 100mg, Pyridoxine 50mg — Single intramuscular dose of hydroxocobalamin 10,000mcg, Thiamin 100mg, Pyridoxine 50mg.
  Other Names: Bedoyecta Tri

SUMMARY:
Demonstrate the effectiveness of a single dose of a multivitamin complex for the treatment of megaloblastic anemia

DETAILED DESCRIPTION:
The investigators will administrate a single intramuscular dose of hydroxocobalamin 10,000mcg, Thiamin 100mg, Pyridoxine 50mg.

To assess response to treatment, a complete blood count (CBC) will be performed weekly during the first month of treatment, after the first month a CBC will be taken monthly for 6 months.

Also to confirm the diagnosis and assess response the investigators will measure levels of methylmalonic acid, homocysteine, and hydroxocobalamin at the beginning of the study, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Age >18, All sex Clinical suspicious of megaloblastic anemia ( cytopenias and macrocytosis (CBC), hypersegmented neutrophils and elevated lactate dehydrogenase) Patients must sign an informed consent indicating that they are aware of the investigational nature of this study -

Exclusion Criteria:

Administration of hydroxocobalamin in the three years before enrollment Patients with active, uncontrolled psychiatric disorders Severe neurologic deficit Known hematologic malignancy Known coagulation disorder that contraindicates intramuscular injection End-stage kidney disease (GFR <15ml/min) Chronic liver disease (Child-Pugh B or C) Pregnant patients Known infection of Hepatitis B or C and HIV Diagnosis of myelodysplastic syndrome

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Hematologic response | 2 month
  Normalization of complete blood count (CBC).
Duration of hematologic response | 6 months
  Duration of response (months) after the administration of megadose of hydroxocobalamin

SECONDARY OUTCOMES:
Measure levels of hydroxocobalamin | Basal, three and six months
Measure levels of methylmalonic acid. | Basal, three and six months
Measure levels of homocysteine. | Basal, three and six months
Evaluate time to hematologic response | 1 month
  Time to response after the administration of 10,000mcg hydroxocobalamin

CONTACTS AND LOCATIONS:
Overall Officials: David Gómez Almaguer, MD, Study Chair — Hospital Universitario Dr. José Eleuterio González
Locations (1):
- Hospital Universitario Dr. Jose E Gonzalez UANL, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
No plans for a sharing plan pre-determined

REFERENCES:
- [Result] Sanz-Cuesta T, Gonzalez-Escobar P, Riesgo-Fuertes R, Garrido-Elustondo S, del Cura-Gonzalez I, Martin-Fernandez J, Escortell-Mayor E, Rodriguez-Salvanes F, Garcia-Solano M, Gonzalez-Gonzalez R, Martin-de la Sierra-San Agustin MA, Olmedo-Luceron C, Sevillano Palmero ML, Mateo-Ruiz C, Medina-Bustillo B, Valdivia-Perez A, Garcia-de Blas-Gonzalez F, Marino-Suarez JE, Rodriguez-Barrientos R, Ariza-Cardiel G, Cabello-Ballesteros LM, Polentinos-Castro E, Rico-Blazquez M, Rodriguez-Monje MT, Soto-Diaz S, Martin-Iglesias S, Rodriguez-Gonzalez R, Breton-Lesmes I, Vicente-Herrero M, Sanchez-Diaz J, Gomez-Gascon T, Drake-Canela M, Asunsolo-del Barco A; OB12 Group. Oral versus intramuscular administration of vitamin B12 for the treatment of patients with vitamin B12 deficiency: a pragmatic, randomised, multicentre, non-inferiority clinical trial undertaken in the primary healthcare setting (Project OB12). BMC Public Health. 2012 May 31;12:394. doi: 10.1186/1471-2458-12-394. PMID 22650964
- [Result] Stabler SP. Vitamin B12 deficiency. N Engl J Med. 2013 May 23;368(21):2041-2. doi: 10.1056/NEJMc1304350. No abstract available. PMID 23697526
- [Result] Green R. Vitamin B12 deficiency from the perspective of a practicing hematologist. Blood. 2017 May 11;129(19):2603-2611. doi: 10.1182/blood-2016-10-569186. Epub 2017 Mar 30. PMID 28360040
- [Result] Sharabi A, Cohen E, Sulkes J, Garty M. Replacement therapy for vitamin B12 deficiency: comparison between the sublingual and oral route. Br J Clin Pharmacol. 2003 Dec;56(6):635-8. doi: 10.1046/j.1365-2125.2003.01907.x. PMID 14616423